CLINICAL TRIAL: NCT01061827
Title: Validation of the French Version of the Geriatric Mental State: a Structured and Standardized Interview for Diagnosis of Psychiatric Disorders in the Elderly
Brief Title: Validation of the French Version of the Geriatric Mental State (GMS)
Acronym: GMS-Package
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: AOHP/04/VC-GMS
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Validate the French Version of GMS Package
Keywords: GMS-package;dementia;depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dementia
- Depression
- Control

SUMMARY:
A major public health issues of today's aging population is the development of knowledge and expertise in geriatric medicine and psychiatry of the elderly. The depressive disorders and dementia, are among the psychiatric conditions most common in older age. They are the subject of much clinical research, in which brain imaging techniques used to establish correlations anatomo-clinical and radiological-clinical. The prerequisite for the realization of such work locally, is the validation in their French version of clinical assessment tools most commonly used internationally, ensuring reliability, acceptability and comparability of results. Among these tools, "Geriatric Mental Schedule (GMS) Package", is the reference tool for research in psychiatry of the elderly. It is a standardized and structured questionnaire that allows to establish with reliability and reproducibility on the basis of answers to questions, major psychiatric diagnoses in the elderly. It has been validated in several languages (German, Spanish, Italian, Dutch, but also Chinese, Korean ...), but is still not available in French.

Hypothesis: Validate the the French version of "Geriatric Mental Schedule (GMS) Package", to establish diagnoses of dementia and depressive disorders.

DETAILED DESCRIPTION:
Patients 65 years or more, Nearest available to assist with the interview of informal caregivers For the subjects in the "dementia", meets the ICD-10 criteria for dementia, and CDR score at 1 to 2, with or without treatment For the subjects in the "depression", ICD-10 criteria for major depression, score on the depression scale MADRS of 18 or more, with or without treatment For control subjects, level of education based on the number of years of schooling (compulsory education until 16 years, extended school) Affiliation with a social security scheme Consent signed by the subject and the near Non-inclusion criteria Subjects with symptoms involving mixed dementia and depression such as not allowing complete ICD-10 criteria for dementia or depression.

ELIGIBILITY:
Inclusion Criteria:

* Nearest available to assist with the interview of informal caregivers For the subjects in the "dementia", meets the ICD-10 criteria for dementia, and CDR score at 1 to 2, with or without treatment For the subjects in the "depression", ICD-10 criteria for major depression, score on the depression scale MADRS of 18 or more, with or without treatment For control subjects, level of education based on the number of years of schooling (compulsory education until 16 years, extended school)

Exclusion Criteria:

* Subjects with symptoms involving mixed dementia and depression such as not allowing complete ICD-10 criteria for dementia or depression.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65 years or more, Nearest available to assist with the interview of informal caregivers For the subjects in the "dementia", meets the ICD-10 criteria for dementia, and CDR score at 1 to 2, with or without treatment For the subjects in the "depression", ICD-10 criteria for major depression, score on the depression scale MADRS of 18 or more, with or without treatment For control subjects, level of education based on the number of years of schooling (compulsory education until 16 years, extended school)
  Non-inclusion criteria Subjects with symptoms involving mixed dementia and depression such as not allowing complete ICD-10 criteria for dementia or depression.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic of dementia and depression | four years
  Validate the French version of the Geriatric Mental State package.The GMS is a standardised, semi-structured interview for examining and recording the mental state in elderly subjects. It allows the classification of patients by symptom profile and can demonstrate changes in profile over time.

SECONDARY OUTCOMES:
Interjudge concordance for discrimination on control,depression and dementia patients | 4 years
  Measure the metrologic qualities, validition,sensibility, specificity against "gold standard" references as MADRS et CDR.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent CAMUS, MD-PHD, Study Director — CHRU TOURS; Philippe NUBUKPO, MD-PHD, Principal Investigator — CHU-Limoges
Locations (2):
- France (2):
  - CHU-Limoges- CMRR, Limoges, Limouzin
  - University Hospital, Tours